CLINICAL TRIAL: NCT05144529
Title: A Randomized Pilot Study to Investigate the Safety and Immunologic Impact of Evolocumab When Given in Combination With Ipilimumab and Nivolumab in Treatment-Naïve Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: A Randomized Pilot Study of Evolocumab Plus Nivolumab/Ipilimumab in Treatment-Naïve Patients With Metastatic NSCLC
Acronym: TOP2101
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scott Antonia (Other)
Responsible Party: Sponsor-Investigator, Scott Antonia, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109594; W81XWH-21-1-0532 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer Metastatic
MeSH Terms: interventions — Nivolumab; Ipilimumab; evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ipilimumab/nivolumab (Active Comparator): Subjects receive ipilimumab 1 mg/kg IV every 6 weeks and nivolumab 240 mg IV every 2 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ipilimumab/nivolumab/evolucumab (Experimental): Subjects receive ipilimumab 1 mg/kg IV every 6 weeks and nivolumab 240 mg IV every 2 weeks plus evolocumab 140 mg SC every 2 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Evolocumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab IV 240 mg
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab IV 1 mg/kg
  Other Names: Yervoy
Drug: Evolocumab — Evolocumab 14 mg subcutaneous injection
  Other Names: Repatha
  Arms: ipilimumab/nivolumab/evolucumab

SUMMARY:
This is a research study to find out the safety and tolerability of combining the drug evolucumab with standard immunotherapy in people with advanced lung cancer (a type called non-small cell lung cancer).

Nivolumab (Opdivo™) and ipilimumab (Yervoy™) are immunotherapy-type drugs which are approved for the treatment of advanced lung cancer that has expression of PD-L1 greater than or equal to 1%. Evolucumab is being combined with nivolumab and ipilimumab to see if it will improve the anti-tumor capabilities of the immunotherapy. Adding evolocumab to the combination of nivolumab and ipilimumab has not been tested in people before and is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have histologically documented or suspected recurrent incurable and/or stage 4 squamous or non-squamous NSCLC.
2. NO prior chemotherapy, radiation therapy or biologic/targeted therapy for current diagnosis recurrent/metastatic NSCLC. Medical therapy (including adjuvant or maintenance immune therapy) for early stage NSCLC allowed if completed > 6 months prior to study enrollment.
3. TPS PD-L1 < 50%
4. Performance Status ECOG 0-1 (Appendix B).
5. Age >18 years old.
6. No active invasive malignancy in the past 2 years other than non-melanoma skin cancer. Cancers that are in-situ are not considered invasive.
7. No autoimmune disease that would constitute contraindication to receive nivolumab
8. Patients must have core needle biopsy tissue that is available and adequate for dedicated research purposes.
9. No excessive risk for CT or ultrasound guided percutaneous biopsy to obtain research biopsy specimen. Risk assessment is to be determined by the treating oncologist and the interventional radiologist.
10. Patients who do not have an indication for a diagnostic biopsy must undergo an elective 'research only' core needle biopsy.
11. Signed written informed consent including HIPAA according to institutional guidelines.
12. Safety laboratory values within institutional normal ranges.

Exclusion Criteria:

* 1) Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.

  2) Has a known history of active TB (Bacillus Tuberculosis) 3) Hypersensitivity to nivolumab or ipilimumab or any of its excipients 4) Hypersensitivity to evolocumab or any of its excipients 5) Patient does not have a site of suspected malignancy that is accessible to pre-treatment biopsy.

  6) Concurrent administration of any other anti-tumor therapy. 7) Has received prior therapy with a PD1, PDL1, or PDL2 inhibitor. 8) Has received therapy with PCSK9 inhibitor within 90 days of study entry. 9) Known active CNS metastases which are symptomatic. Eligible if metastases have been locally treated 14 days prior to cycle 1 day 1, are clinically controlled, and asymptomatic off high dose steroids on cycle 1 day 1(< 2 mg decadron or 10 mg prednisone daily or equivalent allowed). Untreated, asymptomatic brain metastases allowed if subject does not require corticosteroids or anticonvulsant therapy.

  10) Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

  11) Inability to comply with protocol or study procedures. 12) Active infection requiring antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.

  13) Has known history of, or any evidence of active, non-infectious pneumonitis.

  14) Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) 15) Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency etc) is not considered a form of system treatment. Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).

  16) Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity 17) Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

  18) Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

  19) Major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant disorders that in the opinion of the investigator would compromise the safety of the patient of compromise the patient's ability to complete the study.

  20) Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 30 days before or after any dose of nivolumab). Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed. COVID19 vaccines will be allowed on protocol.

  21) Myocardial infarction having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications. Patients with CAD recently treated with surgery and/or stent, if stable without symptomatic angina pectoris, active ischemia are eligible.

  22) Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

  23) Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either psychiatric or physical (e.g., infectious) illness.

  24) Patient takes daily prednisone > 10 mg or the equivalent dose of a different steroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
DLTs | Assessed upon enrollment of first 6 subjects to 30 days after first study dose
  Safety is defined as the incidence of DLTs assessed in the first 6 evaluable subjects
Change in CD3+ tumor infiltrating lymphocytes | Baseline and day 29
  To characterize treatment-related changes in tumor infiltrating lymphocytes (TIL) using immunohistochemistry analysis. The mean and the standard deviation of the pre-treatment CD3+ TILs and the on-treatment CD3+ TILS as well as those of the difference of these ratios will be estimated.

SECONDARY OUTCOMES:
Change in MHC-1 expression | Baseline and day 29
  To assess the change in the degree of surface expression of MHC-I molecules on tumor cells within each patient comparing on-treatment versus pre-treatment biopsy specimens
Progression-free survival (PFS) | Two years
  PFS is defined as the time between initiation of treatment and initial failure (disease progression or death), whichever comes first.
Overall survival (OS) | Two years
  OS is defined as the time from the first dose of study treatment to death.
Objective Response Rate (ORR) | Two years
  Response rate is defined as the proportion of treated subjects with a complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Scott Antonia, MD, Principal Investigator — Duke University
Locations (1):
- Duke Univ. Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT05144529/ICF_000.pdf